CLINICAL TRIAL: NCT07120659
Title: Vacuum Massage vs Tactile Massage for the Treatment of Chronic Neck Pain: A Randomized Controlled Pilot Study Investigating Pain Mechanisms.
Brief Title: Vacuum Massage vs Tactile Massage for the Treatment of Chronic Neck Pain
Acronym: MeCNeck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Frauke Musial, Professor, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Ethics (REK) number 883588; Application 2023-51 (Other: Ekhagastiftelsen)
Record Dates: First submitted 2025-08-04; First posted 2025-08-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain; massage; soft touch massage; vacuum massage; cupping; quantitative sensory testing QST

STUDY DESIGN:
Intervention Model Description: pre-post intervention of two different massage techniques
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intense skin stimulation (Experimental): A vacuum pump provides a type of suction similar to cupping inducing intense manipulation of the skin. The vacuum can be adjusted according to applied suction and air flow.
  The participant will receive 6 therapy sessions of vacuum massage.
  Interventions: Other: vacuum massage
- Light skin stimulation (Active Comparator): Tactile massage (soft touch) is a soft superficial massage which follows the anatomy of the body without penetrating into the deeper tissues.
  The participants will receive 6 therapy sessions.
  Interventions: Other: soft touch massage

INTERVENTIONS:
Other: soft touch massage — Soft superficial massage which follows the anatomy of the body without penetrating into the deeper tissues
  Other Names: tactile massage
  Arms: Light skin stimulation
Other: vacuum massage — Intense stimulation through suction of the skin and deeper layers
  Other Names: cupping massage
  Arms: Intense skin stimulation

SUMMARY:
Chronic pain significantly impacts individuals and society, with about 30% of Norwegian adults affected, making it the leading cause of long-term sick leave and disability benefits. Concerns over addiction to pain medications highlight the need for non-pharmacological treatments, though many such therapies, often complementary or alternative, are not widely available in conventional healthcare. Unclear biomechanisms of these therapies pose challenges for clinical trials and acceptance.

This pilot study aims to explore the effects of two types of massage-cupping massage (CM, intense) and tactile massage (TM, soft)-on chronic neck pain, focusing on their mechanisms of action. Quantitative sensory testing (QST) will be used as a biomarker to assess changes in the pain pathway. A previous feasibility study on CM and QST conducted in Germany informs this research.

The study will recruit 60 patients with chronic neck pain, randomized to CM or TM, with six weekly treatment sessions. QST will be measured before and after treatment to understand therapy-induced changes in the pain pathway. Findings will help tailor massage therapies to individual needs, improve clinical trial quality, and promote the integration of non-pharmacological treatments into conventional care, benefiting a large population in need.

DETAILED DESCRIPTION:
Chronic pain imposes a severe burden for the individuals suffering from it as well as for society. A report from the Norwegian Institute of Public Health from April 2019 summarizes that "Chronic pain affects about 30 per cent of the adult Norwegian population and is the most common reason for long-term sick leave and disability benefit". At the same time there is increasing awareness, that the potential for addiction for some of the pain medications has become a serious public health challenge as well. Thus, there is an urgent need for non-pharmacological interventions, however, most of these interventions belong to the spectrum of complementary and alternative medicine and are often not available through the conventional healthcare system. The fact that the biomechanisms for many of these therapies are unclear, imposes a challenge for the conduction of clinical trials as well as for the acceptance of theses complementary therapies. Thus, the aim of this randomized controlled pilot study is to investigate the effect of massage on chronic neck pain with regard to their mechanism of action. Two types of massage, cupping massage (CM, intense) vs tactile massage (TM, soft) are compared, which differ regarding the intensity of skin receptor stimulation. Quantitative sensory testing (QST) of the pain pathway will be used as a psychophysiological, mechanistic biomarker. Complete QST has rarely been used to evaluate complementary therapies for chronic pain, however a NFR funded feasibility pilot study (case series) on cupping massage and QST has recently been conducted in Jena, Germany, by this group of applicants. The current study will produce pilot data on QST that can be used for sample size estimation in a future clinical trial. A total of n=60 patients with chronic neck pain will be recruited and randomized to either CM or TM. Patients will receive a total of 6 treatment sessions once per week. QST will be measured before and after the treatment. Since QST can describe therapy induced changes in the neuronal pain pathway, it will contribute fundamentally to our understanding of the mechanisms of action of massage and related interventions. This will i) help to tailor massage therapy to the individual needs of patients and thus improve care ii) which will in turn enhance the quality of clinical trials and iii) foster the acceptance of non-pharmacological interventions for the treatment of pain, which may iv) support their integration into conventional care and make these therapies available for the rather large population in need.

ELIGIBILITY:
Inclusion Criteria:

* suffer from non-specific neck pain persisting at least 3 months
* mean pain intensity ≥ 50 on a 0-100 mm visual analogue scale (NRS) with "0" meaning "no pain" and "100" meaning "worst pain imaginable"

Exclusion Criteria:

* neurological symptoms
* having had a vertebral column surgery less than 12 months prior to the study,
* have received TENS, acupuncture, osteopathy, or a chiropractic maneuver or infiltration at the area within 4 weeks prior to the inclusion in the study
* suffer from a congenital deformation of the spine.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | The measurement will take about 2 hours in total; pre and post intervention (5-6 weeks)
  Sensory testing will be performed according to the standard protocol of the German Research Network on Neuropathic Pain (DFNS) and all measurements will be carried out by the same examiner at a defined point of the trapezius muscle on the site with the worst pain, and the foot and the hand as reference areas (norms exist for hand, foot, back and face).

SECONDARY OUTCOMES:
Numerical pain scale | Takes about 20 seconds for the numeric rating scale; pre vs. post intervention (ca. 5-6 weeks)
  ranging from 0="no pain" to 100mm="worst pain imaginable"

OTHER OUTCOMES:
pain diary | 5-6 weeks, 3-5 min / day
  daily characterisation of pain including medication
Neck Disability Index (NDI) | ca 6-10 min before and after the intervention (ca. 5-6 weeks)
  Measures how neck pain has affects the patient's ability to manage in everyday life.
DN4 (Douleur Neuropathique 4) questionnaire | 10 min, before & after intervention (5-6 weeks)
  diagnostic tool used to identify and assess neuropathic pain
SF-36 health survey | ca. 5-10 min, before and after intervention period (5-6 weeks)
  Health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- UiT, The Arctic University of Norway, Institute of Community Medicine, National Research Center in Complementary and Alternative Medicine, NAFKAM, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No
The study is a small pilot study conducted in only one center in Tromso. Thus, there is no need to share individual participant data.